CLINICAL TRIAL: NCT00587041
Title: Use of Oral Probiotics to Reduce Urinary Oxalate Excretion
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); National Center for Research Resources (NCRR) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, John Lieske, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1483-05; R21AT002534 (NIH); UL1RR024150 (NIH); P50DK083007 (NIH)
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Results first posted 2012-05-31 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-04

CONDITIONS: Nephrolithiasis; Hyperoxaluria; Crohn's Disease
Keywords: Synbiotic; Urine Oxalate; Probiotic; Kidney Stone; Gastric Bypass; Crohn's; Stone; Hyperoxaluria; Enteric Hyperoxaluria
MeSH Terms: conditions — Nephrolithiasis; Hyperoxaluria; Crohn Disease; Kidney Calculi; Calculi

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Participants received placebo for 6 weeks: 1 placebo packet daily and 1 placebo capsule twice daily
  Interventions: Other: Placebo
- Oxadrop (Active Comparator): Participants received Oxadrop for 6 weeks: Oxadrop 1 packet daily plus 1 placebo capsule twice daily. Each gram of Oxadrop® contains 2x1011 bacteria (L. acidophilus, L. brevis, S. thermophilus, and B. infantis)
  Interventions: Dietary Supplement: Oxadrop
- Agri-King Synbiotic (Active Comparator): Participants received AKSB for 6 weeks: AKSB 1 capsule twice daily plus 1 placebo packet daily. AKSB contains Fructo-oligosaccharide; Enterococcus faecium (SF68); Saccharomyces cerevisiae subspecies Boulardi; and Saccharomyces cerevisiae
  Interventions: Dietary Supplement: Agri-King Synbiotic (AKSB)

INTERVENTIONS:
Dietary Supplement: Oxadrop — Oxadrop 1 packet daily plus 1 placebo capsule twice daily. Each gram of Oxadrop® contains 2x1011 bacteria (L. acidophilus, L. brevis, S. thermophilus, and B. infantis).
  Arms: Oxadrop
Dietary Supplement: Agri-King Synbiotic (AKSB) — AKSB 1 capsule twice daily plus 1 placebo packet daily. AKSB contains Fructo-oligosaccharide; Enterococcus faecium (SF68); Saccharomyces cerevisiae subspecies Boulardi; and Saccharomyces cerevisiae
  Other Names: AKSB
  Arms: Agri-King Synbiotic
Other: Placebo — 1 placebo packet daily and 1 placebo capsule twice daily
  Arms: Placebo

SUMMARY:
The purpose of this study was to determine the effect of two probiotic preparations (Agri-King Synbiotic and Oxadrop) on urinary oxalate excretion in patients with mild hyperoxaluria. Probiotics are live microorganisms thought to be beneficial to the host organism. Hyperoxaluria is a hereditary disorder that causes a special kind of stone to form in the kidney and urine. Oxalates are naturally-occurring substances found in plants, animals, and in humans. Excretion of oxalates in the urine is a risk factor for kidney stone formation.

Our hypothesis was that the mild hyperoxaluria is due to over absorption of oxalate from food and that probiotics will improve gastrointestinal barrier function to decrease oxalate absorption across the gut (and hence its elimination in the urine).

In the study, participants were randomized to placebo, Agri-King Synbiotic, or Oxadrop, and were treated for 6 weeks. Patients were maintained on a controlled diet to remove the confounding variable of differing oxalate intake and availability from food.

DETAILED DESCRIPTION:
Renal manifestations of chronic hyperoxaluria include nephrolithiasis and, when extreme, interstitial scarring and progressive loss of function. The clinical outcome can be dismal. Although primary hyperoxaluria is relatively rare, hyperoxaluria secondary to gastrointestinal malabsorption is not. Furthermore, the formation of calcium oxalate kidney stones is extremely common, and evidence suggests that minimal, perhaps transient elevations in urinary oxalate concentration may be an important factor in at least a subgroup of these patients with "idiopathic" calcium oxalate urolithiasis. In the case of enteric hyperoxaluria the pathogenic role of oxalate is clear, and renal scarring is commonly observed as a consequence of oxalate exposure and calcium oxalate crystal deposition, in addition to stones. Unfortunately, few satisfactory specific treatments for enteric hyperoxaluria are available. Typical strategies include dietary restriction of oxalate to limit its delivery to the colon; low fat diets to limit malabsorption and distal colonic effects of fatty acids and bile acids; oral calcium to bind oxalate; and bile acid sequestrants like cholestyramine. In its entirety, this regimen is quite rigorous for patients, and even if compliance is achieved the therapy is not always effective. Previous studies have shown that components of the endogenous digestive microflora can utilize oxalate, potentially limiting its absorption from the intestinal lumen. A recent preliminary study demonstrated that a preparation of lactic acid bacteria degraded oxalate in vitro and reduced urinary oxalate excretion when given by mouth. We have recently demonstrated that the same preparation of lactic acid bacilli (Oxadrop) can reduce urinary oxalate excretion in patients with enteric hyperoxaluria. In the current proposal, in a placebo-controlled trial we will determine the effectiveness of this and another probiotic preparation (Agri-King Synbiotic) [AKSB] for the treatment of hyperoxaluria in patients with mild hyperoxaluria, as well as enteric hyperoxaluria.

Specific Aims are: 1) Determine the effect of two probiotic preparations (AKSB and Oxadrop on urinary oxalate excretion in a well-defined group of patients with enteric hyperoxaluria; and 2) Determine the effect of two probiotic preparations (AKSB and Oxadrop) on urinary oxalate excretion in a well-defined group of patients with idiopathic calcium oxalate urolithiasis and mild hyperoxaluria. If results are positive, treatment for calcium oxalate kidney stones could be revolutionized.

ELIGIBILITY:
Inclusion Criteria:

* Enteric hyperoxaluria (>0.5 mM/day; > 45 mg/day) due to fat malabsorption from inflammatory bowel disease (Crohn's Disease). (Patients in remission maintained on stable doses of Remicade/Imuran/Methotrexate every 8 weeks can be recruited as long as the trial can be conducted between 5 and 8 weeks after the last dose); OR
* Enteric hyperoxaluria (>0.5 mM/day; > 45 mg/day) from gastric bypass procedures (gastric bypass for obesity, or other surgical causes of gastric dumping and fat malabsorption (e.g., antrectomy, vagotomy and pyloroplasty for gastric ulcers) (Patients with inflammatory bowel disease must be in clinical remission); OR
* Calcium oxalate nephrolithiasis and mild hyperoxaluria of unknown etiology (>0.35 mM/day) (n=60)
* Presence of radioopaque stones on x-ray, or a history consistent with passage of a stone or stone surgery or extracorporeal shock wave lithotripsy (ESWL) in the last 5 years and if on stone medication, doses have remained stable for at least 3 months
* Stone composition confirmed either by stone analysis demonstrating composition equal to or more than 50% calcium oxalate, or by radiographic demonstration of a calcific renal stone in the presence of hyperoxaluria

Exclusion Criteria:

* On immunosuppressive medications (excluding small stable doses of prednisone of 10 mg or less)
* Human immunodeficiency virus (HIV) infection, known enteric bacterial infection, or history of splenectomy
* Have a current malignancy, other than superficial skin cancers that have been excised, unless they felt to be in complete remission (> 5 years)
* Previous colectomy
* Have completed a course of oral or parenteral antibiotics less than 2 weeks before initiation of the study (patients who require a course of antibiotics during the period of preparation administration will be withdrawn from the study and excluded from the final analysis)
* Patient pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C Lieske, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Lieske JC, Tremaine WJ, De Simone C, O'Connor HM, Li X, Bergstralh EJ, Goldfarb DS. Diet, but not oral probiotics, effectively reduces urinary oxalate excretion and calcium oxalate supersaturation. Kidney Int. 2010 Dec;78(11):1178-85. doi: 10.1038/ki.2010.310. Epub 2010 Aug 25. PMID 20736987

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from Mayo Clinic, Rochester, Minnesota between Mayo 2006 and May 2009.
Period: Overall Study
Arm/Group | Agri-King Synbiotic | Oxadrop | Placebo
Started | 12 | 14 | 14
Completed | 12 | 14 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Agri-King Synbiotic | Oxadrop | Placebo | Total
Number analyzed (Participants) | 12 | 14 | 14 | 40
Age Continuous [Mean (Standard Deviation); unit: years] | 53.65 (17.80) | 54.22 (14.12) | 50.22 (12.79) | 52.79 (14.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2 | 4
  Male | 10 | 14 | 12 | 36
Region of Enrollment [Number; unit: participants]
  United States | 12 | 14 | 14 | 40
Total Kidney Stones Passed [Mean (Standard Deviation); unit: Number of Stones] — Mean number of kidney stones passed prior to study entry
  Number of Stones | 2.36 (2.2) | 1.75 (0.93) | 2.77 (2.35) | 2.25 (1.86)

OUTCOME MEASURES:

1. Primary Outcome: Change in 24-hour Urinary Supersaturation for Calcium Oxalate
Description: Urine is often supersaturated, which favors precipitation of crystalline phases such as calcium oxalate. However, crystals do not always form in supersaturated urine because supersaturation is balanced by crystallization inhibitors that are also present. Supersaturation is calculated by measuring the concentration of all the ions that can interact. Once these concentrations are known, a computer program can calculate the theoretical supersaturation with respect to the important crystalline phases, eg, calcium oxalate. Values for supersaturated ions are expressed in units of Gibbs free energy.
Time Frame: Time zero (on diet but no drug), 6 weeks (on drug and diet)
Population: As urine values for the final visit were not available for 5 subjects, they were not included in the analysis.
Measure: Mean (Standard Deviation); unit: KJoules/mol
Arm/Group | Placebo | Oxadrop | Agri-King Synbiotic
Number analyzed (Participants) | 12 | 13 | 10
KJoules/mol | 1.40 (0.65) | 1.36 (0.67) | 1.42 (0.49)
Statistical Analysis 1: Comparison: Placebo vs Oxadrop vs Agri-King Synbiotic; 80% power for 0.66 DG difference from placebo. The reported value is the overall p-value for CaOx supersaturation by Kruskal-Wallis test of equal change across all three groups, no pair-wise comparison; Test type: Superiority or Other; p = 0.3, Kruskal-Wallis
Statistical Analysis 2: Comparison: Placebo; Ranked sum T-test for placebo group CaOx SS comparison between 0 and 6 weeks; Test type: Superiority or Other; p = 0.045, t-test, 1 sided
Statistical Analysis 3: Comparison: Agri-King Synbiotic; Ranked sum T-test for AKSB group CaOX SS comparison between 0 and 6 weeks; Test type: Superiority or Other; p = 0.67, t-test, 1 sided
Statistical Analysis 4: Comparison: Oxadrop; Ranked-sum T-Test for Oxadrop group CaOX SS comparison between 0 and 6 weeks; Test type: Superiority or Other; p = 0.30, t-test, 1 sided

2. Secondary Outcome: 24 Hour Urine Oxalate Excretion
Description: The amount of oxalate excreted in the urine over a 24 hour period, a risk for calcium oxalate kidney stones
Time Frame: At end of study, approximately 6 weeks
Population: As urine values for the final visit were not available for 5 subjects, they were not included in the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Oxadrop | Agri-King Synbiotic
Number analyzed (Participants) | 12 | 13 | 10
mmol/L | 0.30 (0.10) | 0.31 (0.09) | 0.28 (0.07)

ADVERSE EVENTS:
Time Frame: Subjects were followed for adverse events during the approximate 6 week study period.
Description: Study coordinators called weekly and at the end of the study subjects completed a questionnaire for any adverse events or disease activity.
Arm/Group | Agri-King Synbiotic | Oxadrop | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/12 | 0/14 | 0/14

LIMITATIONS AND CAVEATS:
Small sample size, low oxalate levels in diet

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes